CLINICAL TRIAL: NCT02716298
Title: A Dispensing Clinical of Fanfilcon A Lens Against Lotrafilcon B Lens Over 1 Month Wear Per Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-64
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fanfilcon A (Active Comparator): Study participants are randomized to wear fanfilcon A lens during the crossover study
  Interventions: Device: fanfilcon A
- lotrafilcon B (Active Comparator): Study participants are randomized to wear lotrafilcon B lens during the crossover study.
  Interventions: Device: lotrafilcon B

INTERVENTIONS:
Device: fanfilcon A — contact lens
  Arms: fanfilcon A
Device: lotrafilcon B — contact lens
  Arms: lotrafilcon B

SUMMARY:
This is a study to evaluate the performance of fanfilcon A lens when worn on a daily wear modality over approximately 1 month in comparison to the lotrafilcon B lens.

DETAILED DESCRIPTION:
This is a 45 subject, 1-month dispensing, crossover, double-masked, randomized, bilateral study comparing the test lens against the control lens. Both test and control lenses will be used in a daily wear modality for 1 month each.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Is correctable to a visual acuity of 20/30 or better (in each eye) with their habitual correction and the assigned study lenses;
* Is an adapted soft contact lens wearer (For the purpose of this study: Current lens wear at least 3 days per week, 8 hours each day);
* Demonstrates an acceptable fit with the study lenses.

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Is participating in any concurrent clinical or research study;
* Is a habitual wearer of lotrafilcon B or enfilcon A lenses.
* Has any known active* ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Is pregnant, lactating or planning a pregnancy at the time of enrollment; (by verbal confirmation at the Screening Visit)
* Is aphakic;
* Has undergone refractive error surgery;

  * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, Principal Investigator — Director, Centre for Contact Lens Research
Locations (1):
- Center for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fanfilcon A Then Lotrafilcon B: Study participants are randomized to wear fanfilcon A lens for 1 month, then lotrafilcon B for 1 month during the crossover study
  fanfilcon A: contact lens lotrafilcon B: contact lens
- Lotrafilcon B Then Fanfilcon A: Study participants are randomized to wear lotrafilcon B for 1 month, then fanfilcon A lens for 1 month during the crossover study.
  lotrafilcon B: contact lens fanfilcon A: contact lens
Period: First Intervention (1 Month)
Arm/Group | Fanfilcon A Then Lotrafilcon B | Lotrafilcon B Then Fanfilcon A
Started | 25 | 24
Completed | 24 | 23
Not Completed | 1 | 1
Not completed — Lens discomfort | 1 | 1
Period: Second Intervention (1 Month)
Arm/Group | Fanfilcon A Then Lotrafilcon B | Lotrafilcon B Then Fanfilcon A
Started | 24 | 23
Completed | 24 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Study participants are randomized to wear fanfilcon A lens or lotrafilcon B lens for 1 month during the crossover study
  fanfilcon A: contact lens lotrafilcon B: contact lens
Arm/Group | Overall Participants
Number analyzed (Participants) | 49
Age, Continuous [Mean (Full Range); unit: years] | 27.1 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Subjective Comfort
Description: Subjective ratings on comfort at insertion (at baseline), comfort when lenses are first put in, comfort during the day's wear, and comfort prior to lens removal (1 month) for fanfilcon A and lotrafilcon B lens. (Scale 0-10, 10=Can't feel the lenses, 0=Painful).
Time Frame: Baseline, 1 month
Measure: Median (Standard Deviation); unit: units on a scale
Groups:
- Fanfilcon A: Study participants are randomized to wear fanfilcon A lens for 1 month during the crossover study
  fanfilcon A: contact lens
- Lotrafilcon B: Study participants are randomized to wear lotrafilcon B lens for 1 month during the crossover study.
  lotrafilcon B: contact lens
Arm/Group | Fanfilcon A | Lotrafilcon B
Number analyzed (Participants) | 47 | 47
units on a scale
  Baseline - Comfort at Insertion | 10 (0.93) | 9 (1.83)
  1 Month - Comfort when lenses are first put in | 10 (1.26) | 9 (1.44)
  1 Month - Comfort during the day's wear | 9 (1.32) | 8 (1.53)
  1 Month - Comfort just prior to lens removal | 8 (1.78) | 7 (2.14)

2. Primary Outcome: Subjective Preference
Description: Subjective ratings on preference for fanfilcon A and lotrafilcon B lens. (Strongly prefer fanfilcon A, slightly prefer fanfilcon A, no preference, slightly prefer lotrafilcon B, strongly prefer lotrafilcon B).
  Subject preference in terms of comfort, dryness, clear vision, Lens Handling, digital devices, all day natural comfort, All day comfort, same comfort at the end of the day (EOD), comfortable after the end of 4 weeks, Same comfort at 4 weeks as initial, comfortable in dry environments, help focus effortlessly while using digital devices, help with end of day (EOD) dryness, help eyes feel less tired at EOD (including computer or digital device use), offering clear vision during driving.
Time Frame: 1 month
Measure: Number; unit: percentage of participants
Groups:
- Strongly Prefer Fanfilcon A; Slightly Prefer Fanfilcon A: Study participants are randomized to wear fanfilcon A lens for 1 month during the crossover study
  fanfilcon A: contact lens
- Slightly Prefer Lotrafilcon B; Strongly Prefer Lotrafilcon B: Study participants are randomized to wear lotrafilcon B lens for 1 month during the crossover study
  lotrafilcon B: contact lens
Arm/Group | Strongly Prefer Fanfilcon A | Slightly Prefer Fanfilcon A | No Preference | Slightly Prefer Lotrafilcon B | Strongly Prefer Lotrafilcon B
Number analyzed (Participants) | 47 | 47 | 47 | 47 | 47
percentage of participants
  Comfort | 52 | 16 | 9 | 16 | 7
  Dryness | 43 | 23 | 11 | 14 | 9
  Clear vision | 38.64 | 25.0 | 29.55 | 4.55 | 2.27
  Lens Handling | 9 | 16 | 52 | 23 | 0
  Digital devices | 27.27 | 27.27 | 40.91 | 2.27 | 2.27
  All day natural comfort | 45 | 20 | 14 | 14 | 7
  All day comfort | 27 | 39 | 11 | 18 | 5
  Same comfort at EOD | 41 | 25 | 11 | 14 | 9
  Comfortable after the end of 4 weeks | 50 | 18 | 7 | 20 | 5
  Same comfort at 4 weeks as initial | 43 | 25 | 11 | 14 | 7
  Comfortable in dry environments | 38.64 | 15.91 | 29.55 | 4.55 | 11.36
  Help focus effortlessly while using digital device | 29.55 | 27.27 | 34.09 | 4.55 | 4.55
  Help with EOD dryness | 34 | 25 | 23 | 11 | 7
  Help eyes feel less tired at EOD | 36.36 | 18.18 | 31.82 | 11.36 | 2.27
  Offering clear vision during driving. | 34 | 29 | 26 | 11 | 0

3. Primary Outcome: Lens Wettability
Description: Lens wettability for fanfilcon A and lotrafilcon B lens. (Scale 0-4, 0.25 steps, 0=excellent, 4=severely reduced)
Time Frame: Baseline, 1 month
Population: One participant excluded from analysis at 1 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Lotrafilcon B
Number analyzed (Participants) | 47 | 47
units on a scale
  Baseline | 0.76 (0.61) | 0.56 (0.46)
  1 month: number analyzed (Participants) | 46 | 46
  1 month | 0.85 (0.71) | 1.08 (0.71)

4. Primary Outcome: Surface Deposits
Description: Surface deposits for fanfilcon A and lotrafilcon B lens. (Scale 0-4, 0.25 steps, 0=excellent, 4=severely reduced)
Time Frame: Baseline, 1 month
Population: One participant excluded from analysis at 1 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fanfilcon A | Lotrafilcon B
Number analyzed (Participants) | 47 | 47
units on a scale
  Baseline | 0.14 (0.22) | 0.26 (0.26)
  1 Month: number analyzed (Participants) | 46 | 46
  1 Month | 0.34 (0.45) | 0.41 (0.56)

ADVERSE EVENTS:
Arm/Group | Fanfilcon A | Lotrafilcon B
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other